CLINICAL TRIAL: NCT02330172
Title: Comparison Sugammadex With Neostigmine in Laryngeal Microsurgery.
Brief Title: Sugammadex Provide Better Surgical Condition Compared With Neostigmine in Laryngeal Microsurgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B1312230009
Record Dates: First submitted 2014-12-09; First posted 2015-01-01 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2015-07

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rocuronium 0.45 - neostigmine (Active Comparator): when anesthetic induction, inrocuronium 0.45 mg/kg will be administered for muscle relaxation.
  When the end of operation, a injection of neostigmine or sugammadex will be administered.
  Interventions: Other: Injection of neostigmine or sugammadex
- rocuronium 0.9 - sugammadex (Active Comparator): When anesthetic induction, rocuronium 0.9 mg/kg will be injected to rocuronium 0.9 - sugammadex group for muscle relaxation.
  When the end of operation,, a injection of neostigmine or sugammadex be administered.
  Interventions: Other: Injection of neostigmine or sugammadex

INTERVENTIONS:
Other: Injection of neostigmine or sugammadex — At anesthetic induction, rocuronium 0.45 to rocuronium 0.45 - neostigmine group or rocuronium 0.9 mg/kg to rocuronium 0.9 - sugammadex group will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four (TOF) using nerve stimulator. After operation, neostigmine 50 mcg/kg or sugammadex 4 mg/kgl be injected.
  Other Names: neostigmin or sugammadex

SUMMARY:
This study aims to make a comparison of surgical condition and recovery time between rocuronium 0.45 mg/kg and neostigmine group and rocuronium 0.9 mg/kg and sugammadex group.

DETAILED DESCRIPTION:
This study aims to make a comparison of surgical condition and recovery time between moderate neuromuscular bloackade with reversal using neostigmine group and deep neuromuscular bloackade with reversal using sugammadex group.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist Physical status classification 1 or 2 elective laryngeal microsurgery under general anesthesia

Exclusion Criteria:

* BMI >25 or < 20 kg/m2 Patients taking intercurrent medication Glutamic Oxalacetate Transaminase or Glutamic Pyruvate Transaminase > 40 IU/L, Cr > 1.4 mg/dl

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ah Young Oh, Principal Investigator — Bungdang Seoul National University
Locations (1):
- Eunsu Choi, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi ES, Oh AY, Koo BW, Hwang JW, Han JW, Seo KS, Ahn SH, Jeong WJ. Comparison of reversal with neostigmine of low-dose rocuronium vs. reversal with sugammadex of high-dose rocuronium for a short procedure. Anaesthesia. 2017 Oct;72(10):1185-1190. doi: 10.1111/anae.13894. Epub 2017 May 11. PMID 28493510

RESULTS

PARTICIPANT FLOW:
Groups:
- Rocuronium 0.45 - Neostigmine: when anesthetic induction, inrocuronium 0.45 mg/kg will be administered for muscle relaxation.
  When the end of operation, a injection of neostigmine or sugammadex will be administered.
  Injection of neostigmine or sugammadex: At anesthetic induction, rocuronium 0.45 to rocuronium 0.45 - neostigmine group or rocuronium 0.9 mg/kg to rocuronium 0.9 - sugammadex group will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four (TOF) using nerve stimulator. After operation, neostigmine 50 mcg/kg or sugammadex 4 mg/kgl be injected.
- Rocuronium 0.9 - Sugammadex: When anesthetic induction, rocuronium 0.9 mg/kg will be injected to rocuronium 0.9 - sugammadex group for muscle relaxation.
  When the end of operation,, a injection of neostigmine or sugammadex be administered.
  Injection of neostigmine or sugammadex: At anesthetic induction, rocuronium 0.45 to rocuronium 0.45 - neostigmine group or rocuronium 0.9 mg/kg to rocuronium 0.9 - sugammadex group will be injected for muscle relaxation.
  During surgical procedure, we will monitor train of four (TOF) using nerve stimulator. After operation, neostigmine 50 mcg/kg or sugammadex 4 mg/kgl be injected.
Period: Overall Study
Arm/Group | Rocuronium 0.45 - Neostigmine | Rocuronium 0.9 - Sugammadex
Started | 22 | 22
Completed | 19 | 21
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium 0.45 - Neostigmine | Rocuronium 0.9 - Sugammadex | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants] — From 18 years to 65 years
  Participants
    Population from 18 years to 65 years: <=18 years | 0 | 0 | 0
    Population from 18 years to 65 years: Between 18 and 65 years | 22 | 22 | 44
    Population from 18 years to 65 years: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 16 | 12 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Number of South Korean participants | 22 | 22 | 44
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Laryngoscopic Score
Description: Definitions for evaluation of Laryngoscopycondition.
  : Easy = jaw relaxed, no resistance to blade insertion, fair = jaw not fully relaxed, slight resistance to blade insertion, difficult = poor jaw relaxation, active resistance of the patient to laryngoscopy.
  Variables Excellent Good Poor
Time Frame: At the beginning of surgery, the surgeon rated the laryngoscopy condition
Population: Definitions for evaluation of Laryngoscopycondition.
  : Easy = jaw relaxed, no resistance to blade insertion, fair = jaw not fully relaxed, slight resistance to blade insertion, difficult = poor jaw relaxation, active resistance of the patient to laryngoscopy.
  Variables Excellent Good Poor
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium 0.45 - Neostigmine | Rocuronium 0.9 - Sugammadex
Number analyzed (Participants) | 21 | 19
Participants
  Difficult | 1 | 0
  Fair | 11 | 0
  Easy | 9 | 19
Statistical Analysis 1: Comparison: Rocuronium 0.45 - Neostigmine vs Rocuronium 0.9 - Sugammadex; Test type: Superiority; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Recovery Time From Neuromuscular Blockade
Description: We measured recovery time ffrom the injection of neostigmine or sugammadex to TOF ratio 0.9
Time Frame: from the injection of neostigmine or sugammadex up to 30 minutes
Measure: Mean (Standard Deviation); unit: minute
Arm/Group | Rocuronium 0.45 - Neostigmine | Rocuronium 0.9 - Sugammadex
Number analyzed (Participants) | 21 | 19
minute | 9.9 (4.0) | 2.1 (0.6)
Statistical Analysis 1: Comparison: Rocuronium 0.45 - Neostigmine vs Rocuronium 0.9 - Sugammadex; Test type: Superiority; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: postoperative one month
Description: Adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
  0 means that there were no participants who suffered Adverse events.
Arm/Group | Rocuronium 0.45 - Neostigmine | Rocuronium 0.9 - Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No